CLINICAL TRIAL: NCT03243994
Title: Small Intestinal Absorption in Patients With Chronic Obstructive Pulmonary Disease Complicated by Cor Pulmonale: A Pilot Study
Brief Title: Small Intestinal Absorption in Patients With Chronic Obstructive Pulmonary Disease and Cor Pulmonale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-15019987
Record Dates: First submitted 2017-07-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cor Pulmonale
Keywords: Cor pulmonale; COPD; Malabsorption; D-xylose; Zinc
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Heart Disease; Malabsorption Syndromes

STUDY DESIGN:
Intervention Model Description: All patients had Chronic Obstructive Lung Disease. Those with additional Cor pulmonale was compared to those without
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Experimental): Patients with COPD without Cor Pulmonale
  Interventions: Diagnostic Test: Absorption test with D-xylose and zink
- COPD + Cor Pulmonale (Experimental): Patients with Cor Pulmonale in addition
  Interventions: Diagnostic Test: Absorption test with D-xylose and zink

INTERVENTIONS:
Diagnostic Test: Absorption test with D-xylose and zink — Absorption of D-xylose (25 g) and zinc (132 mg), administered as a single dose. The concentration of D-xylose and zinc was measured in peripheral blood one, two and three hours after ingestion and used as markers of absorption. Furthermore, urine was collected for five hours to determine the amount of excreted D-xylose.

SUMMARY:
Aim: To investigate whether patients with pulmonary hypertension have reduced absorption capacity compared to COPD patients without cor pulmonale potentially due to venous obstruction in the portal vein system.

The presence of cor pulmonale was determined by echocardiography. The concentration of D-xylose and zinc were measured in peripheral blood one, two and three hours after ingestion and used as markers of absorption. Furthermore, urine was collected for five hours to determine the amount of excreted D-xylose.

DETAILED DESCRIPTION:
Background: Cor pulmonale is a common complication to Chronic Obstructive Pulmonary Disease (COPD), and may result in increased pressure in the inferior caval vein and stasis of the liver. The chronic pulmonary hypertension may lead to stasis in the veins from the small intestine and thereby compromise absorption of nutrients.

Aim: To investigate whether patients with pulmonary hypertension have reduced absorption capacity compared to COPD patients without cor pulmonale.

Methods: Absorption of D-xylose (25 g) and zinc (132 mg), administered as a single dose, was tested in 14 COPD patients, seven with and seven without cor pulmonale. The presence of cor pulmonale was determined by echocardiography. The concentration of D-xylose and zinc were measured in peripheral blood one, two and three hours after ingestion and used as markers of absorption. Furthermore, urine was collected for five hours to determine the amount of excreted D-xylose.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD
* Clinically stable = Unchanged medication for COPD for at least 6 months

Exclusion Criteria:

* Unable to understand Danish
* Other clinically important heart-disease than chronic right heart changes presumably due to lung disease
* Clinically significant gastro-intestinal or kidney disease
* Diabetes
* Treatment with corticosteroids for at least 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Absorption fraction of D-xylose | 3 hours
  plasma concentration, mmol/l

SECONDARY OUTCOMES:
Absorption of zinc | 3 hours
  plasma concentration, micromol/l
Absorption fraction of D-xylose | 5 hours
  urine excretion, mmol

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD, MPA, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No
No plans